CLINICAL TRIAL: NCT04003298
Title: Efficacy of the Addition of a Power Interdental Device to an Electric Toothbrush on Gingival Health: a Randomized Controlled Trial.
Brief Title: Efficacy of the Addition of a Power Interdental Device to an Electric Toothbrush on Gingival Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Water Pik, Inc. (Industry)
Collaborators: All Sum Research Center Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26ORWF2019
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Electric toothbrush and power interdental device (Experimental): Electric toothbrush and power interdental device
  Interventions: Device: Electric toothbrush
- Electric toothbrush (Active Comparator): Electric toothbrush
  Interventions: Device: Control

INTERVENTIONS:
Device: Electric toothbrush — Electric toothbrush and power interdental device
  Arms: Electric toothbrush and power interdental device
Device: Control — Oscillating-rotating
  Arms: Electric toothbrush

SUMMARY:
The study is designed to evaluate the clinical changes in gingival health by measuring the reduction of gingival bleeding and inflammation over 4 weeks. Additionally plaque removal will be evaluated after a single use and over 4 weeks.

DETAILED DESCRIPTION:
Data will be analyzed and reported as mean. The target population is approximately 70 healthy adult volunteers. There will be two groups with a total of 35 subjects per group. Subjects will be randomized using a simple random sample. A computer-generated randomization schedule will be prepared by the study statistician. Based on the randomization schedule, patients will be randomly assigned in a 1:1 ratio to receive either:

With 35 subjects per group, the study will have 90% power to detect an average reduction in the percent of sites with BOP of 25%.

The primary outcome will be the reduction in the percentage of sites with bleeding on probing (BOP) after 4 weeks.

Reduction in the percentage of sites with BOP after 2 weeks (+/- 2 days). Reduction in the MGI after 2 (+/- 2 days) and 4 weeks. Reduction in RMNPI Pre & post, 2 weeks and 4 weeks (=/- 2 days)

Data will include whole mouth, approximal, marginal, facial, and lingual analysis for all indices. Intraoral examination will be performed and any adverse events will be reported and followed up.

Subjects will complete a questionnaire at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 70 years of age
* Be able to provide written informed consent prior to participation
* Agree to not participate in any other oral/dental products clinical study for the study duration
* Be in good general health and be a non-smoker
* Have 50% bleeding on probing sites (moderate gingivitis)
* Have no probing depths greater than 4 mm
* Have a minimum of 20 teeth (not including 3rd molars)
* No partial dentures, orthodontic brackets, wires or other appliances
* Agree to refrain from the use of any non-study dental device or oral care product for the study duration
* Agree to return for the scheduled visits and follow study procedures
* Agree to delay dental prophylaxis until study completion
* Have a minimum pre-brushing plaque score of 0.6
* Have a minimum of 1.75 gingivitis score

Exclusion Criteria:

* Have probing depth greater than 4 mm
* Have a systemic disease (ex. Diabetes, autoimmune disease)
* Have advanced periodontitis
* Taking medication that can influence gingival health (ex. Dilantin, Procardia (calcium channel blockers), Cyclosporine, anticoagulants)
* Have orthodontic appliances or removable partial dentures
* Pregnant at time of study
* Use of antibiotics within 6 months of study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Mean change score in bleeding on probing measured at 6 sites per tooth from baseline and between groups at 4 weeks. | 4 weeks
  Bleeding on Probing
Mean change score in gingival inflammation from baseline and between groups measured by Modified Gingival Index at 4 weeks | 4 weeks
  Modified Gingival Index

SECONDARY OUTCOMES:
Mean change score in dental plaque from baseline and between groups measured by Rustogi Modification of the Navy Plaque Index at 4 weeks. | pre & post, 4 weeks
  Rustogi Modification of the Navy Plaque Index

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Qaqish, Study Director — All Sum Research Center Ltd.
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No